CLINICAL TRIAL: NCT01810822
Title: Sex-specific Associations of Variants in the Regulatory Regions of NADPH Oxidase-2 (CYBB) and Gluthatione Peroxidase 4 (GPX4) Genes With Kidney Disease in Type 1 Diabetes.
Brief Title: Sex-specific Association With Kidney Disease
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FMUSP-LIM25-0002
Record Dates: First submitted 2013-03-11; First posted 2013-03-14 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Diabetic Nephropathy
Keywords: oxidative stress; genetic susceptibility; GPX4; NOX2
MeSH Terms: conditions — Diabetic Nephropathies; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Genesis French-Belgium Study: Cross-sectional, multi-center, binational (Belgian and France) study designed to evaluate the genetic components of diabetic nephropathy. It is a cohort with 501 patients, including 279 individuals (55.7%) with diagnosis of diabetic nephropathy.
- GENEDIAB: Cross-sectional, multi-center, binational (Belgian and France) study designed to evaluate the genetic components of diabetic nephropathy. It is a cohort with 444 patients, including 310 individuals (69.8%) with diagnosis of diabetic nephropathy.
- Brazilian cohort: The cohort comprised 451 patients with type 1 diabetes for more than 10 years (56% women; aged 36 ± 11 years, mean ± SD) recruited in diabetes/endocrinology departments of three university hospitals in the cities of São Paulo (SP), Campinas (SP) and Porto Alegre (RS), Brazil.

SUMMARY:
Oxidative stress is involved in the pathophysiology of diabetic nephropathy. The superoxide-generating nicotinamide adenine dinucleotide phosphate-oxidase 2 (NOX2, encoded by the CYBB gene) and the antioxidant enzyme glutathione peroxidase 4 (GPX4) play opposing roles in the balance of cellular redox status. In the present study, we investigated associations of single nucleotide polymorphisms (SNPs) in the regulatory regions of CYBB and GPX4 with kidney disease in patients with type 1 diabetes.

DETAILED DESCRIPTION:
In the present study, three cohorts of type 1 diabetic patients (one Brazilian and two French/Belgium cohorts) were studied for the association with diabetic nephropathy (DN) with a total of 1396 patients. The patients were classified according to the urinary albumin-to-creatinine ratio (ACR) or urinary albumin excretion rate (UAER) in absence of nephropathy, defined as ACR <30 mg/g or UAER < 20 µg/min or < 20 mg/L and plasma creatinine <1.7 mg/dL; incipient nephropathy, defined as persistent microalbuminuria (ACR 30 - 300 mg/g of creatinine or UAER 20 - 200 µg/min or 20 - 200 mg/L) and plasma creatinine <1.7 mg/dL; established diabetic nephropathy, defined as past or present macroalbuminuria (ACR >300 mg/g of creatinine or UAER >200 µg/min or > 200 mg/L) and plasma creatinine <1.7 mg/dL; advanced diabetic nephropathy, defined as past or present macroalbuminuria, plasma creatinine >1.7 mg/dL and any renal replacement therapy. Genotyping of polymorphisms was performed by Real Time PCR using fluorescent-labelled probes.

ELIGIBILITY:
Inclusion Criteria:

* Overt 10 years of Diabetes Mellitus (Brazilian cohort)
* Diagnostic of diabetes before the age of 35 years, with initial ketosis and requirement for permanent insulin treatment within 1 year of diagnosis and past or present diagnosis of diabetic retinopathy. (Genesis cohort).
* Diagnostic of diabetes before the age of 35 years and past or present diagnosis of severe diabetic retinopathy. (GENEDIAB cohort).

Exclusion Criteria:

* Patients presenting autoimmune diseases, HIV or HCV infections (Brazilian cohort)
* Patients with glomerular filtration rate < 60 mL min-1 1.73 m2 without diabetic retinopathy (Brazilian cohort)
* Terminal cancer and personal disability (GENEDIAB cohort).

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Three cohorts pf type 1 diabetic patients were used for the present study. The first one is a Brazilian cohort with 451 patients recruited in diabetes/endocrinology departments of three university hospitals in the cities of São Paulo (SP), Campinas (SP) and Porto Alegre (RS), Brazil between October 2004 and October 2012. The second one is a French/Belgium cohort with 501 patients recruited from both countries between November 1998 to December 2000. The third cohort is a French/Belgium cohort with 444 patients recruited from both countries between May 1994 to April 1995.
Sampling Method: Probability Sample
Enrollment: 1396 (Actual)
Dates: Start 1994-05; Primary Completion 1994-05 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Albumin to Creatinine Ratio | Two Years

CONTACTS AND LOCATIONS:
Overall Officials: Maria L Côrrea-Giannela, Doctor, Study Director — Clinical Hospital/Faculty of Medicine from University of São Paulo; Gilberto Velho, Doctor, Study Director — INSERM U695
Locations (1):
- Faculty of Medicine from University of São Paulo, São Paulo, São Paulo, Brazil